CLINICAL TRIAL: NCT05033132
Title: An Open-label, Multicenter Phase II Study Evaluating Balstilimab Alone or Balstilimab in Combination With Zalifrelimab in Patients With Advanced Cervical Cancer
Brief Title: A Phase II Study of Balstilimab Independently or in Combination With Zalifrelimab in Advanced Cervical Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was never initiated.
Sponsor: Agenus Inc. (Industry)
Collaborators: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-750-CN01
Record Dates: First submitted 2021-08-27; First posted 2021-09-02 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — balstilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Balstilimab (Experimental): Balstilimab monotherapy: approximately 147 patients.
  Interventions: Drug: Balstilimab
- Balstilimab + Zalifrelimab (Experimental): Balstilimab in combination with Zalifrelimab (combination therapy): approximately 30 patients.
  Interventions: Drug: Balstilimab + Zalifrelimab

INTERVENTIONS:
Drug: Balstilimab — Anti-programmed cell death protein 1 (anti-PD-1) monoclonal antibody
  Arms: Balstilimab
Drug: Balstilimab + Zalifrelimab — An anti-PD-1 monoclonal antibody in combination with a cytotoxic T-lymphocyte antigen-4 (CTLA-4) antibody
  Arms: Balstilimab + Zalifrelimab

SUMMARY:
This is an open-label, multi-center Phase II clinical trial to assess the efficacy, safety, and pharmacokinetics of Balstilimab (Treatment Arm 1 - monotherapy) or in combination with Zalifrelimab (Treatment Arm 2 - combination therapy) for treatment of patients with advanced cervical cancer who relapsed or progressed after receiving first-line platinum-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agree to participate by giving written informed consent.
* Diagnosis:

  1. Have a histologically or cytologically confirmed, locally advanced, inoperable and/or metastatic cervical squamous cell carcinoma, cervical adenosquamous cell carcinoma or cervical adenocarcinoma. Note: A pathological report confirmed by histology or cytology of the primary tumor is required for definitive diagnosis. The following cervical tumors are not eligible for inclusion: minimal deviation adenocarcinoma, gastric-type endocervical adenocarcinoma, clear cell adenocarcinoma of the cervix, neuroendocrine carcinoma of the cervix and mesonephric adenocarcinoma.
  2. Patients with recurrent/metastatic cervical cancer who have received at least 1 platinum-based systemic therapy (excluding radiosensitizing chemotherapy) (with or without bevacizumab), and experienced recurrence or progression of cervical cancer or were intolerable to chemotherapy toxicity during or after the systemic therapy and were unable to receive radiotherapy or radical surgery again. Note (definition of failure or intolerability of first-line platinum-based chemotherapy):

     1. Patients with recurrent or metastatic cervical cancer who have experienced disease progression during platinum-based regimen or have experienced disease progression after receiving ≥4 cycles of effective platinum-based regimen (complete response/progressive disease/stable disease) or were intolerable to toxicity caused by platinum during/after platinum-based regimen and were not suitable for continuous platinum-based regimen.

        Or
     2. Patients with cervical cancer progressed or relapsed during neoadjuvant or adjuvant chemotherapy with platinum-based regimen (≥4 cycles if the platinum-based regimen is effective) or within 6 months after the end of the treatment, are deemed to have failed first-line platinum-based chemotherapy.
  3. Programmed death-ligand 1 (PD-L1) positive (combined positive score ≥1).
* Have at least 1 measurable lesion on imaging based on RECIST 1.1. Measurable lesions should have not been treated with topical treatment such as radiotherapy. If the only one measurable lesion has been treated with previous topical treatment (radiotherapy, ablation, vascular intervention, etc.), it is necessary to confirm that the lesion has progressed, otherwise it will be recorded as a non-target lesion.
* Have a life expectancy of at least 3 months.
* Eastern Cooperative Oncology Group performance status of 0 or 1.
* Have satisfactory organ function as indicated by the following laboratory values:

  1. Bone marrow: absolute neutrophil count >1.5 × 10^9/liter (L), platelet count >100 × 10^9/L, and hemoglobin >8 grams (g)/deciliter (80 g/deciliter) (without transfusions of blood or blood component within 2 weeks of test);
  2. Liver: serum total bilirubin (TBIL) level ≤1.5 × upper limit of normal (ULN), aspartate aminotransferase (AST) level ≤2.5 × ULN, alanine aminotransferase (ALT) level ≤2.5 × ULN (TBIL ≤1.5 × ULN, AST ≤5 × ULN, ALT ≤5 × ULN in case of presence of liver metastases);
  3. Serum creatinine ≤1.5 × ULN; or endogenous creatinine clearance ≥50 milliliters/minute for serum creatinine >1.5 × ULN;
  4. Eligible coagulation function, defined as International Normalized Ratio and prothrombin time ≤1.5 x institutional upper limit of normal (IULN); and activated partial thromboplastin time ≤1.5 x IULN.
* No history of other malignancies within 5 years prior to first dose, except for basal cell carcinoma of the skin, superficial bladder cancer, and squamous cell carcinoma of the skin.
* Patient must provide an adequate amount of eligible formalin fixed paraffin-embedded tumor tissue samples, preferably from a recent tumor focus biopsy, or tumor tissue samples collected at or after the diagnosis of advanced or metastatic tumors from the site that has not been previously treated with radiation. If tumor tissue is not available, a tumor biopsy is required.
* Female patients with or without childbearing potential, for the former, the serum pregnancy test should be negative at the time of screening (serum pregnancy test is preferred within 7 days prior to first dose of the investigational drug, otherwise urine pregnancy test is acceptable if serum pregnancy test is not available). Female patients without childbearing potential are defined as follows (for reasons other than medication): ≥45 years of age and menopause for more than 1 year; post hysterectomy, post oophorectomy or post tubal ligation.
* Females of potential pregnancy must use a highly effective method of contraception (e.g., oral contraceptives, intrauterine devices, abstinence or barrier contraception combined with spermicide) throughout the study and continue contraception for 12 months after the end of treatment.
* Is willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigation device within 4 weeks of the first dose of treatment.
* Has an inadequate washout period prior to first dose of study drug defined as: received systemic cytotoxic chemotherapy or biological therapy within 3 weeks before first dose; received radiation therapy within 3 weeks before first dose; experienced major surgical procedures within 4 weeks prior to the first dose.
* Has received prior therapy with any antibody/drug-targeting T-cell co-stimulatory proteins (immune checkpoints), including but not limited to PD-1, PD-L1, CTLA-4, lymphocyte-activation gene 3, therapeutic vaccines, etc.
* Have not recovered from the toxicity of their last systemic antineoplastic therapy to grade 1 or below as defined by National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) 5.0 prior to the first dose of the study. Note: Patients with sensory neuropathy or alopecia grade ≤2 are eligible.
* Is expected to require any other form of systemic or localized antineoplastic therapy while on trial (including maintenance therapy with another agent, radiation therapy, and/or surgical resection).
* Has known severe hypersensitivity reactions to fully human monoclonal antibodies (NCI-CTCAE 5.0 Grade ≥3).
* Received hematopoietic stimulating factor treatment within 14 days (≤14 days) before the first dose of the study drug, such as granulocyte colony-stimulating factor, erythropoietin, etc.
* Central nervous system tumors, brain metastases, or meningeal metastases are found prior to the first dose of the study drug. Note: Patients with brain metastases are eligible for the study when meeting the following requirements: brain metastases prove to be stable (patients are required to provide the most recent head imaging prior to the first dose, with previous head imaging at least 4 weeks apart, for the investigator to determine whether the brain metastases are stable by comparing the results of the two examinations); any neurological symptoms resulting from brain metastases or their treatment must have resolved or be maintainable to a minimal degree and the symptoms can be clinically determined to be sequelae of the treated lesion; brain metastases treated with steroids must not be treated with steroids for at least 4 weeks prior to the first dose.
* Treatment with systemic corticosteroids or any other form of systemic immunosuppression within 7 days (≤7 days) prior to the first dose of the study drug. Note: Combination with corticosteroids for the treatment of immune-related adverse events and prophylactic use of anticontras allergy medications are permitted during the study period; patients requiring daily corticosteroid replacement therapy, e.g., 5 to 7.5 milligrams daily doses of prednisone or equivalent doses of hydrocortisone and steroid therapy (topical, intraocular, intranasal inhalation routes only) may be enrolled in this study. Note: Patients with type 1diabetes, vitiligo, psoriasis, hypothyroidism, or hyperthyroid disease not requiring immunosuppressive treatment are eligible.
* Active autoimmune disease requiring systemic therapy within the past 2 years or history of autoimmune disease or syndrome requiring systemic steroids/immunosuppressive drugs, e.g., hypophysitis, colitis, hepatitis, nephritis, etc. Replacement therapy (e.g., thyroxine, insulin, physiologic corticosteroid replacement therapy for renal or pituitary insufficiency) is not considered systemic immunosuppressive therapy. Note: Patients with type I diabetes, vitiligo, psoriasis, hypo- or hyperthyroidism who do not require immunosuppressive therapy are eligible for the study.
* Has had an allogeneic tissue/solid organ transplant.
* History of interstitial lung disease or a history of pneumonia that has required oral or intravenous corticosteroids.
* Symptoms of an active infection requiring intravenous systemic therapy.
* Positive human immunodeficiency virus antibody or positive syphilis spirochete antibody and positive syphilis spirochete antibody titer test result (i.e., active syphilis infection).
* Presence of active hepatitis B, hepatitis C or tuberculosis. Active hepatitis B and C are defined as follows: active hepatitis B, positive for hepatitis B surface antigen with the hepatitis B virus deoxyribonucleic acid quantification result greater than the ULN; active hepatitis C, positive for hepatitis C antibody with the hepatitis C virus ribonucleic acid quantification result greater than the ULN.
* Has clinically significant (i.e., active) cardiovascular disease. Note: The following cases are observed within 6 months prior to the first dose: heart disease (Class III/IV congestive heart failure or heart block as defined by the New York Heart Association); deep vein thrombosis or pulmonary embolism; myocardial infarction; severe or unstable arrhythmias or angina pectoris; percutaneous coronary intervention, acute coronary syndromes, coronary artery bypass grafting; cerebrovascular accident, transient ischemic attack, cerebral embolism.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
* Has known mental illness that would interfere with compliance with the requirements of the trial.
* Has a history of substance abuse, alcoholism or other addictions.
* Legal incapacity or legal limitation of capacity.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female only
Enrollment: 0 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) Of Balstilimab Monotherapy Per Independent Review Committee (IRC) Assessment Based Upon Response Evaluation Criteria In Solid Tumours (RECIST) 1.1 | 36 months

SECONDARY OUTCOMES:
ORR Of Balstilimab Monotherapy Per Investigator Assessment Based Upon RECIST 1.1 | 36 months
Disease Control Rate (DCR) Of Balstilimab Monotherapy Per IRC And Investigator Assessment Based Upon RECIST 1.1 | 36 months
Duration of Response (DOR) Of Balstilimab Monotherapy Per IRC And Investigator Assessment Based Upon RECIST 1.1 | 36 months
Time to Response (TTR) Of Balstilimab Monotherapy Per IRC And Investigator Assessment Based Upon RECIST 1.1 | 36 months
Progression-free Survival (PFS) Of Balstilimab Monotherapy Per IRC And Investigator Assessment Based Upon RECIST 1.1 | 36 months
Overall Survival (OS) Of Balstilimab Monotherapy Per IRC And Investigator Assessment Based Upon RECIST 1.1 | 48 months
ORR Of Combined Therapy Of Balstilimab And Zalifrelimab Per IRC And Investigator Assessment Based Upon RECIST 1.1 | 36 months
DCR Of Combined Therapy Of Balstilimab And Zalifrelimab Per IRC And Investigator Assessment Based Upon RECIST 1.1 | 36 months
DOR Of Combined Therapy Of Balstilimab And Zalifrelimab Per IRC And Investigator Assessment Based Upon RECIST 1.1 | 36 months
TTR Of Combined Therapy Of Balstilimab And Zalifrelimab Per IRC And Investigator Assessment Based Upon RECIST 1.1 | 36 months
PFS Of Combined Therapy Of Balstilimab and Zalifrelimab Per IRC And Investigator Assessment Based Upon RECIST 1.1 | 36 months
OS Of Combined Therapy of Balstilimab And Zalifrelimab Per IRC And Investigator Assessment Based Upon RECIST 1.1 | 48 months
Peak Plasma Concentration (Cmax) Of Balstilimab And Zalifrelimab | Pre-dose (2 hours prior to dosing [dosing to occur every 6 weeks for up to 24 months/17 cycles or until continued disease progression or intolerable toxicity]), End of Treatment
Time To Peak Plasma Concentration (Tmax) Of Balstilimab And Zalifrelimab | Pre-dose (2 hours prior to dosing [dosing to occur every 6 weeks for up to 24 months/17 cycles or until continued disease progression or intolerable toxicity]), End of Treatment
Half-life (T1/2) Of Balstilimab And Zalifrelimab | Pre-dose (2 hours prior to dosing [dosing to occur every 6 weeks for up to 24 months/17 cycles or until continued disease progression or intolerable toxicity]), End of Treatment
Area Under The Plasma Concentration Versus Time Curve From The Time Of Administration To The Last Measurable Concentration (AUC0-t) Of Balstilimab And Zalifrelimab | Pre-dose (2 hours prior to dosing [dosing to occur every 6 weeks for up to 24 months/17 cycles or until continued disease progression or intolerable toxicity]), End of Treatment
Number Of Participants With Anti-drug Antibodies For Balstilimab And Zalifrelimab | 36 months
Number Of Participants With Treatment-emergent Adverse Events | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Agenus Inc.
Locations (43):
- China (43):
  - Betta Clinical Study Site 4, Bengbu, Anhui
  - Betta Clinical Study Site 2, Hefei, Anhui
  - Betta Clinical Study Site 3, Hefei, Anhui
  - Betta Clinical Study Site 27, Wuhu, Anhui
  - National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, Beijing Municipality
  - Betta Clinical Study Site 25, Beijing, Beijing Municipality
  - Betta Clinical Study Site 42, Chongqing, Chongqing Municipality
  - Betta Clinical Study Site 9, Fuzhou, Fujian
  - Betta Clinical Study Site 22, Xiamen, Fujian
  - Betta Clinical Study Site 41, Lanzhou, Gansu
  - Betta Clinical Study Site 39, Lanzhou, Gansu
  - Betta Clinical Study Site 14, Huizhou, Guangdong
  - Betta Clinical Study Site 18, Meizhou, Guangdong
  - Betta Clinical Study Site 10, Zhanjiang, Guangdong
  - Betta Clinical Study Site 11, Nanning, Guangxi
  - Betta Clinical Study Site 5, Cangzhou, Hebei
  - Betta Clinical Study Site 40, Harbin, Heilongjiang
  - Betta Clinical Study Site 43, Wuhan, Hubei
  - Betta Clinical Study Site 28, Wuhan, Hubei
  - Betta Clinical Study Site 12, Wuhan, Hubei
  - Betta Clinical Study Site 29, Wuhan, Hubei
  - Betta Clinical Study Site 31, Xiangyang, Hubei
  - Betta Clinical Study Site 6, Changde, Hunan
  - Betta Clinical Study Site 36, Changsha, Hunan
  - Betta Clinical Study Site 35, Changsha, Hunan
  - Betta Clinical Study Site 13, Changsha, Hunan
  - Betta Clinical Study Site 21, Nanjing, Jiangsu
  - Betta Clinical Study Site 8, Nanjing, Jiangsu
  - Betta Clinical Study Site 38, Ganzhou, Jiangxi
  - Betta Clinical Study Site 19, Nanchang, Jiangxi
  - Betta Clinical Study Site 20, Nanchang, Jiangxi
  - Betta Clinical Study Site 24, Shangrao, Jiangxi
  - Betta Clinical Study Site 16, Changchun, Jilin
  - Betta Clinical Study Site 15, Changchun, Jilin
  - Betta Clinical Study Site 7, Dalian, Liaoning
  - Betta Clinical Study Site 34, Shenyang, Liaoning
  - Betta Clinical Study Site 17, Shenyang, Liaoning
  - Betta Clinical Study Site 30, Xi'an, Shaanxi
  - Betta Clinical Study Site 23, Taiyuan, Shanxi
  - Betta Clinical Study Site 26, Tianjin, Tianjin Municipality
  - Betta Clinical Study Site 37, Tianjin, Tianjin Municipality
  - Betta Clinical Study Site 32, Ürümqi, Xinjiang
  - Betta Clinical Study Site 33, Hangzhou, Zhejiang